CLINICAL TRIAL: NCT03744065
Title: A Randomized Comparison Between Ultrasound Guided Lumbar Plexus and Suprainguinal Fascia Iliaca Blocks For Total Hip Replacement Analgesia
Brief Title: Lumbar Plexus and Suprainguinal Fascia Iliaca Blocks For Total Hip Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Daniela Bravo Advis, Assistant Professor, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OAIC1001/18
Record Dates: First submitted 2018-11-13; First posted 2018-11-16 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Hip Osteoarthritis; Pain, Acute; Pain, Postoperative; Opioid Use
Keywords: nerve block; fascia iliaca; hip replacement; lumbar plexus
MeSH Terms: conditions — Osteoarthritis, Hip; Acute Pain; Pain, Postoperative

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lumbar plexus block (Active Comparator): Patients randomized to receive an ultrasound-guided lumbar plexus block
  Interventions: Procedure: lumbar plexus block
- Suprainguinal fascia iliaca block (Experimental): Patients randomized to receive an ultrasound-guided suprainguinal fascia iliaca block
  Interventions: Procedure: suprainguinal fascia iliaca block

INTERVENTIONS:
Procedure: lumbar plexus block — Injection with ultrasound guidance of 40 mL of levobupivacaine 0.25% with 5 micrograms of epinephrine per mL and dexamethasone 4 milligrams, in the posteromedial quadrant of psoas muscle
  Arms: Lumbar plexus block
Procedure: suprainguinal fascia iliaca block — Injection with ultrasound guidance of 40 mL of levobupivacaine 0.25% with 5 micrograms of epinephrine per mL and dexamethasone 4 milligrams, underneath the fascia iliaca at the suprainguinal level
  Arms: Suprainguinal fascia iliaca block

SUMMARY:
The nerves from lumbar plexus (LP) are the current target to achieve analgesia after a total hip arthroplasty (THA). Lumbar plexus block (LPB) is an alternative that provides optimal postoperative analgesia. However, many adverse effects and complications have been reported due to its proximity to vital structures. Because of these shortcomings, an alternative to block the LP nerves is required.

In a recent trial suprainguinal Fascia Iliaca Block (SFIB) was reported to provide reliable analgesia in THA. SFIB may carry a lower risk profile, however, no study has compared the efficacy of LPB and SFIB in this setting.

Thus, this randomized trial is set out to compare US guided LPB and SFIB for analgesia after THA. The hypothesis is that both blocks would result in similar postoperative opioid (morphine) consumption at 24 hours and, therefore, designed the study as an equivalence trial.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years
* American Society of Anesthesiologists classification 1-3
* Body mass index between 20 and 35 (kg/m2)

Exclusion Criteria:

* Adults who are unable to give their own consent
* Pre-existing neuropathy (assessed by history and physical examination)
* Coagulopathy (assessed by history and physical examination and, if deemed clinically necessary, by blood work up i.e. platelets ≤ 100, International Normalized Ratio ≥ 1.4 or prothrombin time ≥ 50)
* Renal failure (assessed by history and physical examination and, if deemed clinically necessary, by blood work up i.e. creatinine ≥ 100)
* Hepatic failure (assessed by history and physical examination and, if deemed clinically necessary, by blood work up i.e. transaminases ≥ 100)
* Allergy to local anesthetics (LAs) or morphine
* Pregnancy
* Prior surgery in the corresponding side of the lumbar o suprainguinal area
* Chronic pain syndromes requiring opioid intake at home

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2020-01-22 (Actual); Study Completion 2020-01-23 (Actual)

PRIMARY OUTCOMES:
Morphine consumption over 24 hours | 24 hours post block
  Total morphine consumption over 24 hours post block

SECONDARY OUTCOMES:
Performance time | 2 hours after surgery
  Interval between the start of skin disinfection and the end of local anesthetic injection
Number of needle passes | 2 hours after surgery
  The initial needle insertion counted as the first pass. Any subsequent needle advancement that is preceded by a retraction of at least 10 mm counts as an additional pass
Postoperative static pain at 3 hours after block | 3 hours after the block
  Pain evaluated in Numeric Rating Score from 0 to 10 points
Postoperative static pain at 6 hours after block | 6 hours after the block
  Pain evaluated in Numeric Rating Score from 0 to 10 points
Postoperative static pain at 12 hours after block | 12 hours after the block
  Pain evaluated in Numeric Rating Score from 0 to 10 points
Postoperative static pain at 24 hours after block | 24 hours after the block
  Pain evaluated in Numeric Rating Score from 0 to 10 points
Postoperative dynamic pain at 3 hours after block | 3 hours after the block
  Pain evaluated in Numeric Rating Score from 0 to 10 points
Postoperative dynamic pain at 6 hours after block | 6 hours after the block
  Pain evaluated in Numeric Rating Score from 0 to 10 points
Postoperative dynamic pain at 12 hours after block | 12 hours after the block
  Pain evaluated in Numeric Rating Score from 0 to 10 points
Postoperative dynamic pain at 24 hours after block | 24 hours after the block
  Pain evaluated in Numeric Rating Score from 0 to 10 points
Postoperative static pain at 48 hours after block | 48 hours after the block
  Pain evaluated in Numeric Rating Score from 0 to 10 points
Postoperative dynamic pain at 48 hours after block | 48 hours after the block
  Pain evaluated in Numeric Rating Score from 0 to 10 points
Time until first morphine demand | 48 hours after the block
  Time until first patient-controlled analgesia morphine demand
Block assessment at 3 hours | 3 hours after the block
  Sensorimotor block assessed using a 10-point composite score evaluating sensory block of the lateral femoral cutaneous, femoral and obturator nerves, and motor block of femoral and obturator nerves.
  Sensation will be assessed with ice on then lateral, anterior and medial thigh using a 0 to 2 point scale. 0= no block, patients can feel cold; 1= analgesic block, patient can feel touch but not cold; 2= anesthetic block, patient cannot feel cold or touch.
  Motor function will be assessed for each nerve with a 0 to 2 points scale where 0= no motor block; 1= paresis; 2= paralysis.
Block assessment at 6 hours | 6 hours after the block
  Sensorimotor block assessed using a 10-point composite score evaluating sensory block of the lateral femoral cutaneous, femoral and obturator nerves, and motor block of femoral and obturator nerves.
  Sensation will be assessed with ice on then lateral, anterior and medial thigh using a 0 to 2 point scale. 0= no block, patients can feel cold; 1= analgesic block, patient can feel touch but not cold; 2= anesthetic block, patient cannot feel cold or touch.
  Motor function will be assessed for each nerve with a 0 to 2 points scale where 0= no motor block; 1= paresis; 2= paralysis.
Block assessment at 24 hours | 24 hours after the block
  Sensorimotor block assessed using a 10-point composite score evaluating sensory block of the lateral femoral cutaneous, femoral and obturator nerves, and motor block of femoral and obturator nerves.
  Sensation will be assessed with ice on then lateral, anterior and medial thigh using a 0 to 2 point scale. 0= no block, patients can feel cold; 1= analgesic block, patient can feel touch but not cold; 2= anesthetic block, patient cannot feel cold or touch.
  Motor function will be assessed for each nerve with a 0 to 2 points scale where 0= no motor block; 1= paresis; 2= paralysis.
Incidence of block related adverse events | 3 hours after block
  Incidence of adverse events related to nerve block (vascular puncture, local anesthetic systemic toxicity, epidural spread)
Incidence of opioid related adverse events | 48 hours after block
  Incidence of adverse events related to opioid use (nausea/vomiting, pruritus, somnolence, respiratory depression)
Incidence of Inability to perform physiotherapy | 24 hours after the block
  Inability to perform physiotherapy due to pain (score more than 4 in Numeric Rating Score from 0 to 10 points) or motor blockade.
Surgical duration | 4 hours
  Time between skin incision and closure
Readiness to discharge | 4 days after surgery
  Days to be ready for discharge following physiotherapist criteria
Length of hospital stay | 7 days after surgery
  Length of hospital stay after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Bravo, MD, Principal Investigator — University of Chile
Locations (1):
- Hospital Clínico Universidad de Chile, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siddiqui ZI, Cepeda MS, Denman W, Schumann R, Carr DB. Continuous lumbar plexus block provides improved analgesia with fewer side effects compared with systemic opioids after hip arthroplasty: a randomized controlled trial. Reg Anesth Pain Med. 2007 Sep-Oct;32(5):393-8. doi: 10.1016/j.rapm.2007.04.008. PMID 17961837
- [Background] Klein SM, D'Ercole F, Greengrass RA, Warner DS. Enoxaparin associated with psoas hematoma and lumbar plexopathy after lumbar plexus block. Anesthesiology. 1997 Dec;87(6):1576-9. doi: 10.1097/00000542-199712000-00040. No abstract available. PMID 9416746
- [Background] Aida S, Takahashi H, Shimoji K. Renal subcapsular hematoma after lumbar plexus block. Anesthesiology. 1996 Feb;84(2):452-5. doi: 10.1097/00000542-199602000-00027. No abstract available. PMID 8602680
- [Background] Aveline C, Bonnet F. Delayed retroperitoneal haematoma after failed lumbar plexus block. Br J Anaesth. 2004 Oct;93(4):589-91. doi: 10.1093/bja/aeh242. Epub 2004 Aug 20. PMID 15321930
- [Background] Weller RS, Gerancher JC, Crews JC, Wade KL. Extensive retroperitoneal hematoma without neurologic deficit in two patients who underwent lumbar plexus block and were later anticoagulated. Anesthesiology. 2003 Feb;98(2):581-5. doi: 10.1097/00000542-200302000-00044. No abstract available. PMID 12552223
- [Background] Gentili M, Aveline C, Bonnet F. [Total spinal anesthesia after posterior lumbar plexus block]. Ann Fr Anesth Reanim. 1998;17(7):740-2. doi: 10.1016/s0750-7658(98)80112-3. French. PMID 9750813
- [Background] Pousman RM, Mansoor Z, Sciard D. Total spinal anesthetic after continuous posterior lumbar plexus block. Anesthesiology. 2003 May;98(5):1281-2. doi: 10.1097/00000542-200305000-00034. No abstract available. PMID 12717153
- [Background] Duarte LT, Saraiva RA. [Total spinal block after posterior lumbar plexus blockade: case report.]. Rev Bras Anestesiol. 2006 Oct;56(5):518-23. doi: 10.1590/s0034-70942006000500010. Portuguese. PMID 19468598
- [Background] Dogan Z, Bakan M, Idin K, Esen A, Uslu FB, Ozturk E. Total spinal block after lumbar plexus block: a case report. Braz J Anesthesiol. 2014 Mar-Apr;64(2):121-3. doi: 10.1016/j.bjane.2013.03.002. Epub 2013 Oct 11. PMID 24794455
- [Background] Gadsden JC, Lindenmuth DM, Hadzic A, Xu D, Somasundarum L, Flisinski KA. Lumbar plexus block using high-pressure injection leads to contralateral and epidural spread. Anesthesiology. 2008 Oct;109(4):683-8. doi: 10.1097/ALN.0b013e31818631a7. PMID 18813048
- [Background] Auroy Y, Benhamou D, Bargues L, Ecoffey C, Falissard B, Mercier FJ, Bouaziz H, Samii K. Major complications of regional anesthesia in France: The SOS Regional Anesthesia Hotline Service. Anesthesiology. 2002 Nov;97(5):1274-80. doi: 10.1097/00000542-200211000-00034. PMID 12411815
- [Background] Dalens B, Vanneuville G, Tanguy A. Comparison of the fascia iliaca compartment block with the 3-in-1 block in children. Anesth Analg. 1989 Dec;69(6):705-13. PMID 2589650
- [Background] Dolan J, Williams A, Murney E, Smith M, Kenny GN. Ultrasound guided fascia iliaca block: a comparison with the loss of resistance technique. Reg Anesth Pain Med. 2008 Nov-Dec;33(6):526-31. doi: 10.1016/j.rapm.2008.03.008. PMID 19258967
- [Background] Kumar K, Pandey RK, Bhalla AP, Kashyap L, Garg R, Darlong V, Malhotra R, Yadav CS. Comparison of conventional infrainguinal versus modified proximal suprainguinal approach of Fascia Iliaca Compartment Block for postoperative analgesia in Total Hip Arthroplasty. A prospective randomized study. Acta Anaesthesiol Belg. 2015;66(3):95-100. PMID 26767235
- [Background] Hebbard P, Ivanusic J, Sha S. Ultrasound-guided supra-inguinal fascia iliaca block: a cadaveric evaluation of a novel approach. Anaesthesia. 2011 Apr;66(4):300-5. doi: 10.1111/j.1365-2044.2011.06628.x. Epub 2011 Feb 24. PMID 21401544
- [Background] Desmet M, Vermeylen K, Van Herreweghe I, Carlier L, Soetens F, Lambrecht S, Croes K, Pottel H, Van de Velde M. A Longitudinal Supra-Inguinal Fascia Iliaca Compartment Block Reduces Morphine Consumption After Total Hip Arthroplasty. Reg Anesth Pain Med. 2017 May/Jun;42(3):327-333. doi: 10.1097/AAP.0000000000000543. PMID 28059869
- [Background] Sauter AR, Ullensvang K, Niemi G, Lorentzen HT, Bendtsen TF, Borglum J, Pripp AH, Romundstad L. The Shamrock lumbar plexus block: A dose-finding study. Eur J Anaesthesiol. 2015 Nov;32(11):764-70. doi: 10.1097/EJA.0000000000000265. PMID 26426575
- [Background] Arnuntasupakul V, Chalachewa T, Leurcharusmee P, Tiyaprasertkul W, Finlayson RJ, Tran DQ. Ultrasound with neurostimulation compared with ultrasound guidance alone for lumbar plexus block: A randomised single blinded equivalence trial. Eur J Anaesthesiol. 2018 Mar;35(3):224-230. doi: 10.1097/EJA.0000000000000736. PMID 29135692